CLINICAL TRIAL: NCT01661270
Title: A Multinational, Randomized, Double-Blind Study of Aflibercept Versus Placebo With Irinotecan/ 5-FU Combination (FOLFIRI) in Patients With Metastatic Colorectal Cancer (MCRC) After Failure of an Oxaliplatin Based Regimen
Brief Title: A Study of Aflibercept Versus Placebo With FOLFIRI in Patients With Metastatic Colorectal Cancer Previously Treated With an Oxaliplatin Chemotherapy
Acronym: AFLAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC11338; U1111-1115-7227 (Other: UTN)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo for aflibercept intravenous (IV) infusion on Day 1 of each cycle (1 cycle = 2 weeks) in combination with FOLFIRI regimen until disease progression, unacceptable toxicity or participant's refusal. FOLFIRI regimen: Irinotecan 180 mg/m^2 IV infusion and leucovorin 400 mg/m^2 IV infusion, 5-Fluorouracil IV bolus 400 mg/m^2 followed by continuous IV infusion 2400 mg/m^2.
  Interventions: Drug: Placebo
- Aflibercept (Experimental): Aflibercept 4 mg/kg IV infusion on Day 1 of each cycle (1 cycle = 2 weeks) in combination with FOLFIRI regimen until disease progression, unacceptable toxicity or participant's refusal. FOLFIRI regimen: Irinotecan 180 mg/m^2 IV infusion and leucovorin 400 mg/m^2 IV infusion, 5-Fluorouracil IV bolus 400 mg/m^2 followed by continuous IV infusion 2400 mg/m^2.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Pharmaceutical form: Concentrate for Solution for infusion; Route of administration: Intravenous
  Other Names: AVE0005; Zaltrap
  Arms: Aflibercept
Drug: Placebo — Pharmaceutical form: Concentrate for Solution for infusion; Route of administration: Intravenous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the improvement in progression-free survival (PFS) of aflibercept versus placebo in participants with metastatic colorectal cancer treated with FOLFIRI as second-line treatment for metastatic disease.

Secondary Objectives:

To compare the overall survival (OS) in the 2 treatment arms. To compare the overall response rate (ORR) in the 2 treatment arms. To assess the safety profile of the 2 treatment arms. To assess immunogenicity of intravenous (IV) aflibercept in selected centers.

DETAILED DESCRIPTION:
Screening occurred from signed informed consent to randomization (up to 21 days). A treatment cycle was defined as a 2 week-period. All participants were followed during the study treatment and follow-up period until death or study cut off date, which ever comes first.

ELIGIBILITY:
Inclusion criteria:

* Histological or cytological proven adenocarcinoma of the colon or rectum.
* Metastatic disease that was not amenable to potentially curative treatment.
* One and only one prior chemotherapeutic regimen for metastatic disease. This prior chemotherapy must be an oxaliplatin containing regimen. Participants who were relapsed within 6 months of completion of oxaliplatin based adjuvant chemotherapy were eligible.

Exclusion criteria:

* Prior therapy with irinotecan.
* Eastern Cooperative Oncology Group (ECOG) performance status >1.
* Less than 28 days elapsed from prior radiotherapy, from prior surgery and prior chemotherapy to the time of randomization. Less than 42 days elapsed from prior major surgery to the time to randomization.
* Adverse events (with exception of alopecia, peripheral sensory neuropathy grade ≤ 2 and those listed in specific exclusion criteria) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.3.0) at the time of randomization.
* Age <18 years.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Other prior malignancy. Adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or any other cancer from which the participants had disease free for > 5 years were allowed.
* Participation in another clinical trial with an investigational drug and any concurrent treatment with any investigational drug within 30 days prior to randomization.
* Any of the following within 6 months prior to randomization: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association Functional Classification (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior to randomization: treatment resistant peptic or duodenal ulcer disease, erosive oesophagitis or gastritis, grade 3 or 4 gastrointestinal bleeding/hemorrhage, gastrointestinal perforation/fistula, abdominal abscess, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
* Participants who had given high dose of aspirin or non steroidal anti-inflammatory agents (NSAIDS) or high steroids within 4 weeks prior to randomization. The definition of "high dose" was to be based on the investigator's judgment.
* Occurrence of deep vein thrombosis within 4 weeks, prior to randomization.
* Inadequate organ or bone marrow function.
* Pregnant or breast-feeding woman. Positive serum or urine pregnancy test prior to randomization. Participants with reproductive (M/F) who were not agree to use accepted and effective method of contraception during the study treatment period and for at least 6 months following completion of study treatment.
* Uncontrolled hypertension.
* Urine Protein: creatine ratio (UPCR) >1 on morning spot urinalysis or proteinuria > 500mg/24 hours.
* Participants on anticoagulant therapy with unstable dose of warfarin and/or having an out-of-therapeutic range international normalized ratio (INR) (>3) within 4 weeks prior to randomization.
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy.
* Known dihydropyrimidine dehydrogenase deficiency.
* Predisposing colonic or small bowel disorder in which the symptoms were uncontrolled as indicated by baseline of > 3 loose stools daily.
* Prior history of chronic enteropathy, inflammatory enteropathy, chronic diarrhea, unresolved bowel obstruction/sub-obstruction, more than hemicolectomy, extensive small intestine resection with chronic diarrhea.
* History of anaphylaxis or known intolerance to atropine sulphate or loperamide or appropriate antiemetics to be administered in conjunction with FOLFIRI.
* Treatment with concomitant anticonvulsant agents that were cytochrome P450 3A4 (CYP3A4) inducers (phenytoin, phenobarbital, carbamazepine), unless discontinued > 7 days.
* Participants with known Gilbert's syndrome.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- China (21):
  - Investigational Site Number 156003, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156004, Beijing
  - Investigational Site Number 156016, Chengdu
  - Investigational Site Number 156020, Chongqing
  - Investigational Site Number 156021, Fuzhou
  - Investigational Site Number 156008, Guangzhou
  - Investigational Site Number 156010, Hangzhou
  - Investigational Site Number 156011, Hangzhou
  - Investigational Site Number 156009, Hangzhou
  - Investigational Site Number 156015, Harbin
  - Investigational Site Number 156012, Nanjing
  - Investigational Site Number 156013, Nanjing
  - Investigational Site Number 156006, Shanghai
  - Investigational Site Number 156007, Shanghai
  - Investigational Site Number 156014, Shenyang
  - Investigational Site Number 156005, Tianjin
  - Investigational Site Number 156019, Wuhan
  - Investigational Site Number 156018, Wuhan
  - Investigational Site Number 156017, Xi'an
- Hong Kong (2):
  - Investigational Site Number 344002, Hong Kong
  - Investigational Site Number 344001, Shatin, Nt
- Japan (10):
  - Investigational Site Number 392006, Amagasaki-Shi
  - Investigational Site Number 392003, Bunkyō City
  - Investigational Site Number 392004, Bunkyō City
  - Investigational Site Number 392009, Gifu
  - Investigational Site Number 392002, Kitaadachi-Gun
  - Investigational Site Number 392001, Kobe
  - Investigational Site Number 392005, Kochi
  - Investigational Site Number 392007, Kumamoto
  - Investigational Site Number 392008, Nagakute-Shi
  - Investigational Site Number 392010, Takatsuki-Shi
- Singapore (2):
  - Investigational Site Number 702002, Singapore
  - Investigational Site Number 702001, Singapore
- Taiwan (2):
  - Investigational Site Number 158003, Taipai
  - Investigational Site Number 158002, Taipei

REFERENCES:
- [Derived] Li J, Xu R, Qin S, Liu T, Pan H, Xu J, Bi F, Lim R, Zhang S, Ba Y, Bai Y, Fan N, Tsuji A, Yeh KH, Ma B, Wei V, Shi D, Magherini E, Shen L. Aflibercept plus FOLFIRI in Asian patients with pretreated metastatic colorectal cancer: a randomized Phase III study. Future Oncol. 2018 Aug;14(20):2031-2044. doi: 10.2217/fon-2017-0669. Epub 2018 Aug 17. PMID 30117334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 37 centers in 5 countries. A total of 332 participants were randomized between 17 July 2012 and 18 March 2014.
Pre-assignment Details: Due to treatment kit misallocation, part of the patients randomized to placebo received aflibercept for
  1/several treatment cycles and are presented as a separate group for safety evaluation.
  EOT criteria were: disease progression/death, un-tolerable toxicity, consent withdrawal/Investigator decision.
Period: Overall Study
Arm/Group | Placebo | Aflibercept
Started | 109 | 223
Adverse Event | 26 (Met end of treatment (EOT) criteria.) | 47 (Met EOT criteria)
Disease Progression | 67 (Met EOT criteria) | 118 (Met EOT criteria)
Physician Decision | 1 (Met EOT criteria) | 8 (Met EOT criteria)
Participant's Request | 15 (Met EOT criteria) | 48 (Met EOT criteria)
Other Reasons | 0 | 2
Completed | 109 (Treatment until disease progression/death, toxicity, consent withdrawal or Investigator's decision.) | 223 (Treatment until disease progression/death, toxicity, consent withdrawal or Investigator's decision.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo for IV infusion on Day 1 of each cycle (1 cycle = 2 weeks) in combination with FOLFIRI regimen until disease progression, unacceptable toxicity or participant's refusal. FOLFIRI regimen: Irinotecan 180 mg/m^2 IV infusion and leucovorin 400 mg/m^2 IV infusion, 5-Fluorouracil IV bolus 400 mg/m^2 followed by continuous IV infusion 2400 mg/m^2.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aflibercept | Total
Number analyzed (Participants) | 109 | 223 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (11.3) | 55.1 (10.9) | 54.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 95 | 141
  Male | 63 | 128 | 191

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time interval from the date of randomization to the date of first observation of either tumor progression or death due to any cause. Tumor assessment was performed by Independent Review Committee (IRC) as per response evaluation criteria in solid tumors (RECIST) version 1.0. Progression was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study or absolute increase and at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was calculated by Kaplan-Meier estimates.
Time Frame: 26.7 months
Population: Intent-to-Treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 109 | 223
months | 5.59 [4.632 to 6.111] | 6.93 [6.045 to 7.655]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the earliest between the last date of the participants was known to be alive and the study cut-off date. Analysis was performed by Kaplan-Meier method.
Time Frame: 31.6 months
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 109 | 233
months | 11.93 [10.086 to 14.292] | 14.59 [13.175 to 16.460]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate was defined as the proportion of participants with confirmed complete response (CR) or confirmed partial response (PR), as assessed by Investigators and the IRC according to RECIST 1.0 criteria, relative to the total number of participants in the relevant analysis population. Complete Response (CR): disappearance of all target and non-target lesions and no new lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions with no progression of non-target lesions and no new lesions, or, the disappearance of all target lesions but persistence of 1 or more non-target lesions not qualifying for either CR or progressive disease (PD) and no new lesions.
Time Frame: 26.6 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 109 | 233
percentage of participants | 3.7 [NA to NA] — Insufficient number of participants for the CI to be calculated | 18.4 [13.3 to 23.5]

ADVERSE EVENTS:
Time Frame: All AE collected from signature of informed consent upto resolution/stabilization/death regardless of seriousness/relationship to IMP.After cutoff date for OS,only ongoing AE & SAE were followed until resolution,stabilization/2 follow-ups(about 4 months).
Description: Reported AEs were treatment-emergent AEs that developed/worsened during 'on-treatment period' (from first dose of Aflibercept to 30 days of follow-up visit). Safety population (subset of ITT population): all participants who received at least one dose of study drug. Due to operational treatment error, 3 arms were reported for safety analysis.
Groups:
- Placebo Only: Placebo for IV infusion on Day 1 of each cycle (1 cycle = 2 weeks) in combination with FOLFIRI regimen until disease progression, unacceptable toxicity or participant's refusal. FOLFIRI regimen: Irinotecan 180 mg/m^2 IV infusion and leucovorin 400 mg/m^2 IV infusion, 5-Fluorouracil IV bolus 400 mg/m^2 followed by continuous IV infusion 2400 mg/m^2.
- Aflibercept Only: Aflibercept 4 mg/kg IV infusion on Day 1 of each cycle (1 cycle = 2 weeks) in combination with FOLFIRI regimen until disease progression, unacceptable toxicity or participant's refusal. FOLFIRI regimen: Irinotecan 180 mg/m^2 IV infusion and leucovorin 400 mg/m^2 IV infusion, 5-Fluorouracil IV bolus 400 mg/m^2 followed by continuous IV infusion 2400 mg/m^2.
- Mixed Administration (Placebo and Aflibercept): Participants who were originally randomized to receive either Placebo or Aflibercept, actually received both the treatment (Placebo and Aflibercept).
Arm/Group | Placebo Only | Aflibercept Only | Mixed Administration (Placebo and Aflibercept)
Serious Adverse Events (participants affected / at risk) | 9/33 | 30/111 | 43/188
Other Adverse Events (participants affected / at risk) | 32/33 | 109/111 | 188/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Only (N=33) | Aflibercept Only (N=111) | Mixed Administration (Placebo and Aflibercept) (N=188)
Anal abscess (Infections and infestations) | 1 | 1 | 3
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 1
Catheter site abscess (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 3
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 2
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2 | 5
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Only (N=33) | Aflibercept Only (N=111) | Mixed Administration (Placebo and Aflibercept) (N=188)
Upper respiratory tract infection (Infections and infestations) | 1 | 11 | 19
Urinary tract infection (Infections and infestations) | 0 | 3 | 14
Neutropenia (Blood and lymphatic system disorders) | 22 | 68 | 135
Leukopenia (Blood and lymphatic system disorders) | 20 | 59 | 84
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 22 | 24
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 12
Decreased appetite (Metabolism and nutrition disorders) | 15 | 42 | 90
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 15 | 11
Insomnia (Psychiatric disorders) | 4 | 9 | 10
Headache (Nervous system disorders) | 1 | 9 | 17
Dizziness (Nervous system disorders) | 4 | 8 | 17
Cholinergic syndrome (Nervous system disorders) | 4 | 7 | 11
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 4
Hypertension (Vascular disorders) | 1 | 43 | 65
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 30 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 13 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 11
Nausea (Gastrointestinal disorders) | 22 | 61 | 110
Diarrhoea (Gastrointestinal disorders) | 14 | 60 | 122
Vomiting (Gastrointestinal disorders) | 22 | 56 | 107
Stomatitis (Gastrointestinal disorders) | 5 | 27 | 60
Abdominal pain (Gastrointestinal disorders) | 4 | 19 | 42
Constipation (Gastrointestinal disorders) | 8 | 14 | 35
Abdominal distension (Gastrointestinal disorders) | 4 | 13 | 11
Mouth ulceration (Gastrointestinal disorders) | 2 | 11 | 29
Abdominal pain upper (Gastrointestinal disorders) | 0 | 7 | 15
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 6 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 6 | 3
Toothache (Gastrointestinal disorders) | 2 | 2 | 2
Rectal discharge (Gastrointestinal disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 9 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 8 | 10
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 8 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5 | 43
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 5 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 14
Proteinuria (Renal and urinary disorders) | 0 | 19 | 37
Haematuria (Renal and urinary disorders) | 1 | 6 | 5
Fatigue (General disorders) | 9 | 37 | 84
Pyrexia (General disorders) | 3 | 15 | 33
Asthenia (General disorders) | 1 | 12 | 24
Chest discomfort (General disorders) | 2 | 2 | 4
Pain (General disorders) | 2 | 1 | 5
Alanine aminotransferase increased (Investigations) | 2 | 11 | 19
Weight decreased (Investigations) | 1 | 9 | 27
Aspartate aminotransferase increased (Investigations) | 2 | 8 | 21
Blood pressure increased (Investigations) | 0 | 8 | 6
White blood cell count decreased (Investigations) | 3 | 7 | 16
Haemoglobin decreased (Investigations) | 1 | 5 | 15
Platelet count decreased (Investigations) | 2 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.